CLINICAL TRIAL: NCT05047965
Title: Evaluation of MRI With Dixon Based Sequences in the Detection of Prostate Cancer
Brief Title: An Investigational Scan (MRI With Dixon Based Sequences) in Detecting Prostate Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-0003; NCI-2019-02461 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0003 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (standard MRI, Dixon MRI) (Experimental): Patients undergo MRI with additional Dixon based sequences with fat and water over a total of 49 minutes.
  Interventions: Procedure: Dixon MRI; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Dixon MRI — Undergo Dixon MRI
  Other Names: Dixon Fat-Suppression MRI
Procedure: Magnetic Resonance Imaging — Undergo standard MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This trial studies the use of magnetic resonance imaging (MRI) with Dixon based imaging sequences in detecting prostate cancer. MRI uses radio waves and a powerful magnet linked to a computer to create detailed pictures of areas inside the body. Researchers hope to learn if using a modified MRI scan technique with Dixon based imaging sequencing will help to produce better images of prostate cancer than the standard of care MRI scan technique.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate prospectively the accuracy of Dixon based sequences in detection of intraprostatic tumor nodules.

II. Determine the sensitivity, specificity, positive and negative predictive value of Dixon based sequences in assessment of extraprostatic tumor extension and lymph node involvement.

SECONDARY OBJECTIVES:

I. Compare the accuracy of Dixon based sequences versus multiparametric diffusion weighted imaging including diffusion tensor imaging in tumor detection and extraprostatic extension.

II. Compare the accuracy of Dixon based sequences in detection of transition zone tumors.

III. Determine the optimal scanning parameters for Dixon based sequences in the imaging of prostate adenocarcinoma.

OUTLINE:

Patients undergo MRI with additional Dixon based sequences with fat and water over a total of 49 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate cancer patients who are scheduled to undergo prostatectomy.
* Patient who is scheduled to have a clinically indicated staging endorectal prostate MRI exam.
* Patients who have signed their informed consent form to undergo the study.

Exclusion Criteria:

* Known prior hormone ablation or radiation therapy (pelvic or prostate).
* Patients who do not want to undergo prostatectomy and prefer other therapy or surveillance.
* Contraindication to conventional MR imaging (e. g. metal implants, pace maker, etc.).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2013-04-25 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Detection of at least one or more prostate lesions with Dixon sequencing | through study completion, an average of 1 year
  Will evaluate and compare the accuracy of Dixon based sequencing to the conventional T2 weighted sequencing for detection of intraprostatic tumor and extraprostatic tumor extension. Lesions will be within any of six regions of the prostate: left apex, left mid, left base, right apex, right mid, and right base. The relative sensitivity and specificity of the two sequencing methods will be compared using an adjusted McNemar's test for clustered data where clusters consist of the matched pairs of within patient-zone observations. The primary analysis will also provide 95% confidence intervals for marginal sensitivity and specificity using a generalized linear mixed model.

CONTACTS AND LOCATIONS:
Overall Officials: Ganeshan Dhakshina Moorthy, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org